CLINICAL TRIAL: NCT05561855
Title: The Effect of mHealth-Based Lifestyle Intervention on Overweight or Obese Patients With Type 2 Diabetes: A Randomized Controlled Trial
Brief Title: T2DM Intensity Lifestyle Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo No. 1 Hospital (Other)
Collaborators: Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NBFH20220755
Record Dates: First submitted 2022-09-22; First posted 2022-09-30 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus, Type 2; Overweight or Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lifestyle intervention (Experimental): 1. Weight monitoring: Participants are required to record the weighting data in the WeChat official account at least once a week to lose 5% or more of their initial body weight in 3 months.
  2. Goals record: At baseline, the participants need to complete a behavioral goals questionnaire. All these behaviors are then ranked for each participant based on an algorithm that determines the participants'self-reported necessity, self-efficacy, and estimated caloric deficit from performing that behavior. The top six goals are assigned to each participant with two for every 4-week cycle.
  3. Exercise: The form is the combination of aerobic exercise (3d/w) and resistance exercise(2d/w). Each participant will be equipped with a Huami watch as a means of monitoring.
  4. Health education: Participants are provided with T2DM-related knowledge. They can also contact the endocrinologist online and offline.
  Interventions: Behavioral: lifestyle intervention
- usual-care control (No Intervention): Participants assigned to the control group will receive routine medical care and diabetes education, and be treated with hypoglycemic drugs under the guidance of endocrinologists according to the patient's condition and clinical treatment standards throughout their participation in the trial. After finishing the study, they will be offered healthy management as the participants in the multi-component lifestyle intervention group.

INTERVENTIONS:
Behavioral: lifestyle intervention — During the 3-month lifestyle intervention period, the participants need to complete the weight monitoring, behavioral goal recording, diet and exercise recording, online course learning by using the WeChat official account module of "Weight Loss and Glucose Control".They will receive corresponding feedback and integral rewards every week, and receive monthly follow-ups to complete health education, goal review, motivational interview as well as collecting medication changes and blood glucose monitoring data.
  Arms: lifestyle intervention

SUMMARY:
This RCT study will evaluate the effect of a lifestyle intervention on overweight or obese patients with type 2 diabetes mellitus. The primary hypothesis is that the mHealth-based intensive lifestyle intervention is sufficient to achieve weight loss and maintain glycated hemoglobin control.

DETAILED DESCRIPTION:
Diabetes mellitus is a chronic systemic metabolic disease caused by the long-term interaction of genetic factors and environmental factors. It is characterized by an increase in plasma glucose levels and is mainly due to metabolic disorders in glucose, fat, and protein caused by insufficient insulin secretion and/or dysfunction in the body, which affects normal physiological activities. As of 2019, 463 million people are suffering from diabetes in the world, of which 90% to 95% have type 2 diabetes mellitus (T2DM), with an average of 1 patient in every 11 adults (aged 20-79). The number of patients with T2DM will jump to 700 million by 2045. There is a close relationship between T2DM and overweight and obesity. The prevalence of diabetes in overweight and obese people in China was 12.8% and 18.5%, respectively. Among T2DM patients, the proportions of overweight and obesity were 41% and 24.3%, respectively.The two kinds of diseases share a common key pathophysiological mechanism, which will have a devastating long-term impact on patients' health and bring serious disease and economic burden to the family. Given the various harms, it is urgent to carry out relevant intervention research and formulate effective intervention strategies. With the development of artificial intelligence technology, the combination of mHealth and multidisciplinary lifestyle intervention may become an efficient and easy-to-popularize management mode for the prevention and treatment of T2DM with obesity.

Given the relative lack of high-quality interventions for T2DM overweight/obesity, the investigators designed a randomized controlled trial to assess the effectiveness of a multicomponent intervention in Ningbo First Hospital. This study plans to adopt the online and offline combination method based on mHealth technology to carry out lifestyle intervention aimed at formulating a set of feasible and effective intervention strategies.

The study aims to identify: 1) whether the mHealth-based intensive lifestyle intervention will be effective for weight and glycated hemoglobin management to reverse or slow down the disease process among T2DM patients with overweight/obesity; 2) whether the intervention will be beneficial for improving biochemical indicators, body composition indicators, and exercise capacity among T2DM patients with overweight/obesity.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the WHO diagnostic criteria for type 2 diabetes;
2. The duration of diabetes is less than 5 years;
3. HbA1c was between 6.5-11% in recent 3 months;
4. 18-65 years old;
5. 24kg/m2≤BMI#40kg/m2;
6. Weight loss within the past 3 months did not exceed 5% of initial weight;
7. Currently using a smartphone;
8. Voluntary participation.

Exclusion Criteria:

1. Pregnant or lactating woman, or planning a pregnancy within 6 months after recruitment;
2. Uncontrolled hypertension (resting blood pressure ≥ 160/100mmHg);
3. Treatment with insulin;
4. Acute complications of diabetes (diabetic ketoacidosis, hyperosmolar state, infection. etc) have occurred within the past 3 months, or one or more severe chronic complications of diabetes have existed, such as severe cardiovascular or cerebrovascular pathology (angina pectoris, myocardial infarction, grade III-IV heart failure, severe arrhythmia, transient cerebral ischemic attack, stroke, etc.), massive proteinuria (urinary albumin/creatinine ratio ≥300 mg/g), and severe diabetic foot, severe neuropathy, blurred vision.
5. Currently using weight-reducing products such as orlistat, or other medications that can significantly affect weight such as diuretics and hormones;
6. Severe cardiovascular and cerebrovascular diseases, respiratory diseases, hepatic and renal insufficiency, malignant tumors and other chronic consumptive diseases, active infections, and surgical history involving important organs within 3 months;
7. Contraindications to physical activity;
8. The presence of mental or cognitive impairment;
9. Current participation in other clinical trial projects;
10. Having the same family member involved in the research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Weight change from baseline | at end of the 3-month intervention
  measured in kilograms (kg) and calculate the change percentage(%)
The change of HbA1c from baseline | at end of the 3-month intervention
  measured in percent (%)

SECONDARY OUTCOMES:
The change in body mass index (BMI) from baseline | at end of the 3-month intervention
  Weight and height will be combined to report BMI in kg/m^2.
The change of waist circumference from baseline | at end of the 3-month intervention
  measured in centimetre (cm)
The change of waist-to-hip circumference ratio from baseline | at end of the 3-month intervention
  measure waist circumference and hip circumference to calculate waist-to-hip circumference ratio
The change of both systolic and diastolic blood pressures from baseline | at end of the 3-month intervention
  measure systolic and diastolic blood pressure in millimeters of mercury (mmHg) by using electronic sphygmomanometer
The change of body fat percentage from baseline | at end of the 3-month intervention
  measure body fat percentage (%) by bioelectrical impedance analysis
The change of blood lipids from baseline | at end of the 3-month intervention
  measure total cholesterol, triglyceride, high-density lipoprotein cholesterol, and low-density lipoprotein cholesterol in milligram/deciliter (mg/dL)
The change in muscle strength from baseline | at end of the 3-month intervention
  measure grip strength in kilograms (kg) by hand dynamometer
The change in exercise capacity from baseline | at end of the 3-month intervention
  The 3-Minute Step Test is an assessment for Cardiorespiratory Fitness. At the end of the 3 minutes, sit down and monitor the pulse for one full minute. Calculate step-test index with the recovery heart rate. The fitter you are, the quicker the heart rate will return to normal after exercise.
The change in life quality from baseline | at end of the 3-month intervention
  It is measured in the form of the Short form health survey (SF-36), scored from 0 to 100, with higher scores associated with better quality of life.
The change in sleep quality from baseline | at end of the 3-month intervention
  It is measured in the form of the Pittsburgh Sleep Quality Index (PSQI), scored from 0 to 21, with higher scores associated with worse quality of sleep.
The change in depression severity from baseline | at end of the 3-month intervention
  It is measured in the form of the Pittsburgh Sleep Quality Index (PSQI), scored from 0 to 27, with higher scores associated with greater degree of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Li Li, Bachelor, Principal Investigator — Ningbo No. 1 Hospital
Locations (1):
- Ningbo First Hospital, Ningbo, Zhejiang, China